CLINICAL TRIAL: NCT05529524
Title: Signatures of Response and Resistance to Mosunetuzomab in Follicular Lymphomas (FL)
Status: Completed | Type: Observational
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: CALC
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Follicular Lymphoma
Keywords: Follicular Lymphoma; Mosunetuzomab; Resistance; CD20-CD3; Bispecific antibodies; Neoplasms; Lymphatic Diseases; Immunoproliferative Disorders
MeSH Terms: conditions — Lymphoma, Follicular; Neoplasms; Lymphatic Diseases; Immunoproliferative Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Lymph node biopsies: Cryostor, Formalin-Fixed, Paraffin-Embedded (FFPE), and frozen
  * Whole blood
  * Bone marrow aspiration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mosunetuzumab is a T-cell bispecific antibody targeting CD20 and CD3 aiming to redirect T cells to engage and eliminate malignant B cells. Bispecific antibodies (BsAb) are a promising treatment option which can induce long-term responses in refractory and relapsed B cell lymphoma patients. However, the factors determining the quality and duration of responses are poorly understood.

DETAILED DESCRIPTION:
the objective is to produce a collection of great scientific interest for lymphoma research from CELESTIMO's clinical trial patients' samples to increase knowledge of treatment with mosunetuzumab's for patients with follicular lymphoma (FL).

study population involves patients participating to CELESTIMO study in France. 10 sites are expected in this biobanking protocol study

Biological samples will collected as part of routine care (tissue and blood already sampled in routine and/or CELESTIMO study) at screening, at C4, at C12 or at progressive disease/relapse.

ELIGIBILITY:
patients who participate to CELESTIMO study (NCT04712097)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who participate to CELESTIMO study (NCT04712097)
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Capacity of sampling | 2 years
  number of samples collected

CONTACTS AND LOCATIONS:
Overall Officials: Camille Laurent, MD, Principal Investigator — Oncopole - Toulouse France; Karin Tarte, PhD, Principal Investigator — Micro-environnement et cancer (MICA) - Rennes France; Franck MORSCHHAUSER, MD, Principal Investigator — Centre Hospitalier Universitaire de Lille - Lille France
Locations (9):
- France (9):
  - Centre Hospitalier de La Cote Basque; Hematologie, Bayonne
  - Hopital Claude Huriez; Hematologie, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU Saint Eloi; Service d'Hématologie Clinique, Montpellier
  - CHU NANTES - Hôtel Dieu; Service d'Hematologie Clinique, Nantes
  - CHU de Nîmes - Hôpital Carémeau, Nîmes
  - Hopital Saint Antoine; Hematologie Clinique, Paris
  - Hopital De La Miletrie; Hematologie Et Oncologie Medicale, Poitiers
  - CHU Pontchaillou, Rennes

IPD SHARING:
Plan to Share IPD: No